CLINICAL TRIAL: NCT06755411
Title: Oral Health Promotion and Fundamental of Care: an Evidence-based Practice Educational Program
Brief Title: Oral Health and Fundamental of Care Program
Acronym: OHFCP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Dal Molin (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Sponsor-Investigator, Alberto Dal Molin, PhD, Associate Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Organization: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CE078/2023
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Oral Hygiene, Oral Health; Oral Cavity; Nursing Care; Nursing Education
Keywords: oral hygiene; oral health; fundamental of care; nursing care; nursing education

STUDY DESIGN:
Intervention Model Description: Study design: the effectiveness of an evidence-based practice educational program to improve the quality of oral care has been evaluated in a before-and-after quasi-experimental study.
  The study adhered to The TREND statement guidelines, which provide a 22-item checklist designed to ensure consistent reporting of nonrandomized controlled trials. This statement, which is complementary to the widely recognized CONSORT statement for randomized controlled trials, was utilized to guide the study's methodology (Des Jarlais, Lyles, Crepaz, & TREND Group, 2004).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-intervention group (No Intervention): The pre-intervention group was recruited between May and June 2023. At admission, every 5 days, and at discharge, an expert (dentists and/or dental hygienists) inspected the patient's oral cavity. The specialist personnel of the Department of Dentistry recorded data and observations on the proper documentation approved by the local ethics committee, combining the collection of socio-demographic data with the completion of the OHAT scale through its Italian validated version and the Internal Protocol of the Surgical Department of Dentistry (standard protocol). The expert panel assessed the selected patients during the following time frame: T0a (at admission); T0d (at discharge); T0i 1, 2, 3,… (intermediate) at five-day intervals until discharge, always at the same ideal time (about 9.00 am). Data collection required approximately 15 minutes per patient each time.
- OHFCP2 (Active Comparator): The intervention consists of a two-phase approach for implementing guidelines and evidence-based recommendations: educating healthcare professionals and enhancing clinical activity. A training course was developed for nurses and social health professionals. Lecture sessions on the most recent literature were held, as well as practical learning training sessions in high fidelity simulation, which included the assessment, preservation, and care of the oral and dental health.The intervention was administered to small groups consisting of 5-6 participants. An in-patient room situation with three possible scenarios and corresponding simulation manikins was set up: a person with a healthy oral cavity, a person with prosthesis, and an edentulous old person. After implementing the educational intervention, a new data collection phase began in the same hospital department during December replicating the same patient recruitment and evaluation process.
  Interventions: Other: OHFCP2

INTERVENTIONS:
Other: OHFCP2 — The proposed intervention consists of a two-phase approach for implementing guidelines and evidence-based recommendations: educating healthcare professionals and enhancing clinical activity.
  Arms: OHFCP2

SUMMARY:
Introduction:

Oral health significantly impacts daily life, affecting communication, nutrition, emotional expression, self-esteem, and overall quality of life. Poor oral health is associated with conditions ranging from caries and periodontal disease to systemic issues such as diabetes, cardiovascular disorders, and increased mortality.

Background and Rationale:

Oral frailty, a concept originating in Japan in 2013, highlights the deterioration of oral function due to aging, potentially leading to malnutrition and systemic health impacts. The 2017 Global Burden of Disease Study emphasized oral health as an ongoing global challenge, identifying caries, severe periodontitis, and edentulism as prevalent issues. Preventable oral diseases contribute significantly to health disparities and systemic illnesses.

Aims:

Primary: To evaluate the impact of an educational intervention to implement evidence-based guidelines for oral health care in adult inpatients.

Secondary: To assess the concordance between different assessment tools and the improvement in knowledge of healthcare workers following training.

Methods:

Study Design: A before-and-after interventional study comparing pre- and post-educational intervention implementation cohorts.

Setting: Medical Department, Maggiore della Carità Hospital, Novara, Italy. Eligibility: Adults aged ≥18 years admitted for inpatient care who consent to participate.

Outcomes: Improvements in oral health outcomes as assessed by the OHAT tool and secondary metrics such as knowledge improvement in healthcare staff.

Intervention:

Training Sessions: Healthcare workers receive education on oral health guidelines, including practical and simulation-based activities.

Implementation: Adoption of evidence-based practices for oral health care.

Evaluation Phases:

Phase 1 (Baseline): Assessment of oral health in patients using OHAT and a structured evaluation protocol.

Phase 2 (Intervention): Educational sessions for healthcare workers. Phase 3 (Post-Implementation): Follow-up assessments using the same tools and methods as Phase 1.

Data Analysis:

Statistical methods include descriptive analysis, repeated measures models, and pre-post intervention comparisons. A significance level of 0.05 will be applied.

Sample Size:

A minimum of 48 participants (24 per cohort) is required, based on a hypothesised effect size of 0.5 with 80% power and a significance level of 0.05.

Ethical Considerations:

The protocol will be submitted for ethical approval. Data will be anonymised and handled per EU Regulation 2016/679 (GDPR).

Dissemination of Results:

Findings will be published in peer-reviewed journals and presented at conferences, maintaining participant confidentiality.

DETAILED DESCRIPTION:
Background Oral health care encompasses all practices of education, motivation, prevention, assessment, and care delivery aimed at preventing and/or eliminating soft and hard tissue pathologies within the oral cavity or slowing their progression.

The literature highlights that oral hygiene needs are often not addressed at the same level as other health needs, and certain populations are at a higher risk of poor oral health compared to others.

Providing effective oral hygiene is essential to ensuring both local and systemic well-being. Oral health education aims to enhance knowledge and skills while promoting good practices to reduce morbidity associated with the oral cavity. Conversely, a lack of education and training strategies, as well as failure to implement preventive measures, inevitably leads to a progressive increase in oral health issues.

In the context of person-centered care, the standards derived from the delivery of fundamental care represent the baseline below which care quality should not fall. These standards are supported by robust evidence and defined through Clinical Practice Guidelines (CPGs).

Based on these considerations, a before-and-after study was designed to evaluate the effectiveness of an evidence-based guideline implementation program for oral health care and management, targeting nursing staff and healthcare assistants in the Internal Medicine Ward of the AOU Maggiore della Carità, Novara.

Global and Local Context The Global Burden of Disease Study 2017 provided a global perspective on the prevalence, incidence, and disability-adjusted life expectancy associated with oral health conditions, stratified by age, gender, and country from 1990 to 2017. The results demonstrate that oral health conditions and their management remain a significant global challenge.

Worldwide, oral health pathologies affect 3.5 billion individuals, including:

2.4 billion with untreated caries in permanent teeth (35% of the global population).

796 million with severe periodontitis. 532 million with untreated caries in primary teeth. 267 million with total edentulism. 139 million with other pathological conditions.

Oral cancer is among the top three cancers in the Pacific region of Asia. Most oral health conditions are preventable, can be intercepted early, and treated effectively. Notably, there is a well-established correlation between proper oral care and systemic conditions such as cardiovascular disorders, hypertension, stroke, diabetes, dementia, respiratory diseases, and increased mortality.

Assessment Tools for Oral Health Various tools are available to assess oral health status or estimate risks. The Registered Nurses' Association of Ontario (RNAO) recommends standardized approaches or validated tools for comprehensive assessment of oral and peri-oral structures, including evaluation of breath, hygiene, and pain.

The Oral Health Assessment Tool (OHAT), tested in various settings for adults, is practical, reliable, and quick for use by non-specialized healthcare staff. A validated Italian version is also available.

Study Objective This before-and-after study aims to assess the impact of implementing evidence-based guidelines for oral health care among adult patients admitted to a medical ward, focusing on changes in oral health-related outcomes.

Secondary Objectives:

Estimate concordance between adopted assessment tools. Evaluate changes in healthcare staff's knowledge of guidelines and best practices for oral health care.

Methodology Data collection will follow specific time points: upon admission, every five days, and at discharge. Assessments will include the OHAT scale and a protocol tailored for specialized oral health evaluations.

Primary Outcome: oral health improvement assessed using OHAT. Secondary Outcomes: Concordance between OHAT and standard protocol tailored for specialized oral health evaluations.

Knowledge improvement among staff pre- and post-training.

Intervention Phases

1. Baseline Evaluation (T0): Oral health assessment using OHAT and per standard protocol upon admission, intermediate days, and discharge.
2. Training Program: Implementation of RNAO guidelines in two stages:

   Healthcare Staff Education Clinical workflow restructuring.
3. Post-Implementation Evaluation (T1): Reassessment using the same tools.

Sample Size and Statistical Analysis A minimum of 24 patients per group is required to detect an effect size of 0.5 with 80% power at a 0.05 significance level. Statistical analysis will compare changes in OHAT scores between groups using repeated measures models, chi-square tests, or non-parametric equivalents as appropriate.

Ethical Considerations The protocol will be submitted to the Institutional Ethics Committee for approval. Participants will provide informed consent, and data will be handled anonymously in compliance with GDPR regulations. Any protocol amendments will be reported promptly.

Conclusion This study seeks to provide evidence for the effectiveness of training programs and guideline implementation in improving oral health care practices, ultimately benefiting patient outcomes both locally and systemically.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the requirements for the study should have been at least 18 years old, be admitted on a regular schedule, and be able to understand and give informed consent for the study. Patients assigned, even temporarily, to other inpatient wards were not eligible
* Only patients admitted to Internal General Medicine Ward at Maggiore della Carità Hospital, Novara, a 640-bed university hospital in northern Italy.

Exclusion Criteria:

* Patients unable to understand and consent, with critical conditions preventing oral cavity assessment (e.g., presence of non-removable non-invasive ventilatory support devices, transient disorientation, unwillingness to participate) were excluded. Patients had the right to withdraw their participation agreement at any point during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Variation of OHAT score related to educational intervention and timing T0, T5 and T100 (discharge) | T0= ADMISSION; T5= DAY-5 (and every 5-days until discharge); T=100 (discharge)
  The Oral Health Assessment Tool (OHAT) uses a Likert scale ranging from 0 (very healthy) to 2 (very unhealthy) for each item, with a total of 8 items assessed. The maximum score is 16, and higher scores indicate worse oral health conditions.
  The OHAT average score differences in the pre-post-intervention phases, assessing if the educational intervention produces an effect of reducing the progression of oral cavity deterioration. Regarding the analysis of mouth conditions, any changes between admission and discharge were assessed with the OHAT tool. Because the data are correlated (evaluated at separate times) and classified into three groups (good, sufficient, and inadequate) Bhapkar's test was applied. The same assessment was done assuming that just the difference between T5 and T100 is reported, excluding the first evaluation upon admission, because it is influenced by oral hygiene practices carried out at home or in other setting.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Gallione, PhD, MSN, RN, Principal Investigator — AOU Maggiore della Carità di Novara; Cristian Vairo, PhD st, MSN, RN, Study Chair — AOU Maggiore della Carità di Novara
Locations (1):
- AOU Maggiore della Carità, Novara, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu, J.-H., Liu, M., Ho, M.-H., & Chang, C.-C. (2017). Oral Health of Older Adults in Long-Term Care Facilities: Effects of an Oral Care Program. J Oral Health Dent Care, 1(2), 1:008.
- [Background] Wong FMF, Shie HWH, Kao E, Tsoi HM, Leung WK. Educational Programme on Knowledge, Attitudes, and Practice of Oral Care/Hygiene Provision by Healthcare Providers to Older Residents in Long-Term Care Institutions: A Case-Control Study. Geriatrics (Basel). 2024 Jan 29;9(1):16. doi: 10.3390/geriatrics9010016. PMID 38392103
- [Background] WHO. (2020). World Health Organization. Retrieved Nov. 2020, from Home/Health topics/Oral health: https://www.who.int/health-topics/oral-health/#tab=tab_1
- [Background] Spoon D, Rietbergen T, Huis A, Heinen M, van Dijk M, van Bodegom-Vos L, Ista E. Implementation strategies used to implement nursing guidelines in daily practice: A systematic review. Int J Nurs Stud. 2020 Nov;111:103748. doi: 10.1016/j.ijnurstu.2020.103748. Epub 2020 Aug 18. PMID 32961463
- [Background] Sist L, Contini C, Bandini A, Bandini S, Massa L, Zanin R, Maricchio R, Gianesini G, Bassi E, Tartaglini D, Palese A, Ferraresi A. [MISSCARE Survey - Italian Version: findings from an Italian validation study]. Ig Sanita Pubbl. 2017 Jan-Feb;73(1):29-45. Italian. PMID 28428643
- [Background] Sasso L, Bagnasco A, Zanini M, Catania G, Aleo G, Santullo A, Spandonaro F, Icardi G, Watson R, Sermeus W. The general results of the RN4CAST survey in Italy. J Adv Nurs. 2017 Sep;73(9):2028-2030. doi: 10.1111/jan.13066. Epub 2016 Jul 26. No abstract available. PMID 27399267
- [Background] Sabbah W, Folayan MO, El Tantawi M. The Link between Oral and General Health. Int J Dent. 2019 May 29;2019:7862923. doi: 10.1155/2019/7862923. eCollection 2019. No abstract available. PMID 31275387
- [Background] Rootman I, Goodstadt M, Potvin L, Springett J. A framework for health promotion evaluation. WHO Reg Publ Eur Ser. 2001;(92):7-38. No abstract available. PMID 11729789
- [Background] RNAO. (2020, May). Registered Nurses Association of Ontario (RNAO). Retrieved 2023 Mar, from Best practice guidelines: https://rnao.ca/bpg/guidelines/oral-health-supporting-adults-who-require-assistance-second-edition
- [Background] RNAO. (2020). Oral Health: Supporting Adults Who Require Assistance, Second Edition. In R. N. l'Ontario (Ed.), Best Practice Guideline. International Affairs and Best Practice Guideline (BPG) Oral Health .
- [Background] RNAO. (2008). Oral Health: Nursing Assessment and Interventions. Nursing Best Practice Guideline. Toronto: Registered Nurses' Association of Ontario.
- [Background] Razak PA, Richard KM, Thankachan RP, Hafiz KA, Kumar KN, Sameer KM. Geriatric oral health: a review article. J Int Oral Health. 2014 Nov-Dec;6(6):110-6. PMID 25628498
- [Background] Prendergast V, Kleiman C, King M. The Bedside Oral Exam and the Barrow Oral Care Protocol: translating evidence-based oral care into practice. Intensive Crit Care Nurs. 2013 Oct;29(5):282-90. doi: 10.1016/j.iccn.2013.04.001. Epub 2013 May 20. PMID 23702324
- [Background] Petersen PE, Baez RJ, Ogawa H. Global application of oral disease prevention and health promotion as measured 10 years after the 2007 World Health Assembly statement on oral health. Community Dent Oral Epidemiol. 2020 Aug;48(4):338-348. doi: 10.1111/cdoe.12538. Epub 2020 May 8. PMID 32383537
- [Background] Peres MA, Macpherson LMD, Weyant RJ, Daly B, Venturelli R, Mathur MR, Listl S, Celeste RK, Guarnizo-Herreno CC, Kearns C, Benzian H, Allison P, Watt RG. Oral diseases: a global public health challenge. Lancet. 2019 Jul 20;394(10194):249-260. doi: 10.1016/S0140-6736(19)31146-8. PMID 31327369
- [Background] NICE. (2016, Dec 15). Oral health promotion in the community. Retrieved Mar 2021, from National Institute for Health and Care Excellence: https://www.nice.org.uk/guidance/qs139
- [Background] NICE. (2016, July 5). Oral health for adults in care homes. Retrieved Mar 2023, from National Institute for Health and Care Excellence: www.nice.org.uk/guidance/ng48
- [Background] NICE. (2014, October 22). Oral health: local authorities and partners. Retrieved Mar 2023, from National Institute for Health and Care Excellence: https://www.nice.org.uk/guidance/ph55
- [Background] NICE. (2012). How NICE clinical guidelines are developed: an overview for stakeholders, the public and the NHS. (N. I. Excellence, Ed.)
- [Background] Ni Chroinin D, Montalto A, Jahromi S, Ingham N, Beveridge A, Foltyn P. Oral Health Status Is Associated with Common Medical Comorbidities in Older Hospital Inpatients. J Am Geriatr Soc. 2016 Aug;64(8):1696-700. doi: 10.1111/jgs.14247. Epub 2016 Aug 3. PMID 27487009
- [Background] National Institute of Dental and Craniofacial Research. (2018, Jul.). Tooth Loss. Retrieved Nov. 2020, from NHI: https://www.nidcr.nih.gov/research/data-statistics/tooth-loss/seniors
- [Background] Moher D, Schulz KF, Altman DG; CONSORT GROUP (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. Ann Intern Med. 2001 Apr 17;134(8):657-62. doi: 10.7326/0003-4819-134-8-200104170-00011. PMID 11304106
- [Background] Malengreaux S, Doumont D, Scheen B, Van Durme T, Aujoulat I. Realist evaluation of health promotion interventions: a scoping review. Health Promot Int. 2022 Oct 1;37(5):daac136. doi: 10.1093/heapro/daac136. PMID 36166263
- [Background] Maeda K, Mori N. Poor oral health and mortality in geriatric patients admitted to an acute hospital: an observational study. BMC Geriatr. 2020 Jan 28;20(1):26. doi: 10.1186/s12877-020-1429-z. PMID 31992227
- [Background] Lugtenberg M, Zegers-van Schaick JM, Westert GP, Burgers JS. Why don't physicians adhere to guideline recommendations in practice? An analysis of barriers among Dutch general practitioners. Implement Sci. 2009 Aug 12;4:54. doi: 10.1186/1748-5908-4-54. PMID 19674440
- [Background] Liao YM, Tsai JR, Chou FH. The effectiveness of an oral health care program for preventing ventilator-associated pneumonia. Nurs Crit Care. 2015 Mar;20(2):89-97. doi: 10.1111/nicc.12037. Epub 2014 Dec 23. PMID 25532600
- [Background] Kossioni AE, Hajto-Bryk J, Janssens B, Maggi S, Marchini L, McKenna G, Muller F, Petrovic M, Roller-Wirnsberger RE, Schimmel M, van der Putten GJ, Vanobbergen J, Zarzecka J. Practical Guidelines for Physicians in Promoting Oral Health in Frail Older Adults. J Am Med Dir Assoc. 2018 Dec;19(12):1039-1046. doi: 10.1016/j.jamda.2018.10.007. PMID 30471798
- [Background] Kim J, Park JH, Shin S. Effectiveness of simulation-based nursing education depending on fidelity: a meta-analysis. BMC Med Educ. 2016 May 23;16:152. doi: 10.1186/s12909-016-0672-7. PMID 27215280
- [Background] Kemppainen V, Tossavainen K, Turunen H. Nurses' roles in health promotion practice: an integrative review. Health Promot Int. 2013 Dec;28(4):490-501. doi: 10.1093/heapro/das034. Epub 2012 Aug 10. PMID 22888155
- [Background] Kalisch BJ, Landstrom GL, Hinshaw AS. Missed nursing care: a concept analysis. J Adv Nurs. 2009 Jul;65(7):1509-17. doi: 10.1111/j.1365-2648.2009.05027.x. Epub 2009 May 9. PMID 19456994
- [Background] Jones TL, Hamilton P, Murry N. Unfinished nursing care, missed care, and implicitly rationed care: State of the science review. Int J Nurs Stud. 2015 Jun;52(6):1121-37. doi: 10.1016/j.ijnurstu.2015.02.012. Epub 2015 Feb 23. PMID 25794946
- [Background] Haghighi A, Shafipour V, Bagheri-Nesami M, Gholipour Baradari A, Yazdani Charati J. The impact of oral care on oral health status and prevention of ventilator-associated pneumonia in critically ill patients. Aust Crit Care. 2017 Mar;30(2):69-73. doi: 10.1016/j.aucc.2016.07.002. Epub 2016 Aug 4. PMID 27499527
- [Background] Institute of Medicine (US) Committee on Standards for Developing Trustworthy Clinical Practice Guidelines; Graham R, Mancher M, Miller Wolman D, Greenfield S, Steinberg E, editors. Clinical Practice Guidelines We Can Trust. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209539/ PMID 24983061
- [Background] GBD 2017 Oral Disorders Collaborators; Bernabe E, Marcenes W, Hernandez CR, Bailey J, Abreu LG, Alipour V, Amini S, Arabloo J, Arefi Z, Arora A, Ayanore MA, Barnighausen TW, Bijani A, Cho DY, Chu DT, Crowe CS, Demoz GT, Demsie DG, Dibaji Forooshani ZS, Du M, El Tantawi M, Fischer F, Folayan MO, Futran ND, Geramo YCD, Haj-Mirzaian A, Hariyani N, Hasanzadeh A, Hassanipour S, Hay SI, Hole MK, Hostiuc S, Ilic MD, James SL, Kalhor R, Kemmer L, Keramati M, Khader YS, Kisa S, Kisa A, Koyanagi A, Lalloo R, Le Nguyen Q, London SD, Manohar ND, Massenburg BB, Mathur MR, Meles HG, Mestrovic T, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mokdad AH, Morrison SD, Nazari J, Nguyen TH, Nguyen CT, Nixon MR, Olagunju TO, Pakshir K, Pathak M, Rabiee N, Rafiei A, Ramezanzadeh K, Rios-Blancas MJ, Roro EM, Sabour S, Samy AM, Sawhney M, Schwendicke F, Shaahmadi F, Shaikh MA, Stein C, Tovani-Palone MR, Tran BX, Unnikrishnan B, Vu GT, Vukovic A, Warouw TSS, Zaidi Z, Zhang ZJ, Kassebaum NJ. Global, Regional, and National Levels and Trends in Burden of Oral Conditions from 1990 to 2017: A Systematic Analysis for the Global Burden of Disease 2017 Study. J Dent Res. 2020 Apr;99(4):362-373. doi: 10.1177/0022034520908533. Epub 2020 Mar 2. PMID 32122215
- [Background] Gostemeyer G, Baker SR, Schwendicke F. Barriers and facilitators for provision of oral health care in dependent older people: a systematic review. Clin Oral Investig. 2019 Mar;23(3):979-993. doi: 10.1007/s00784-019-02812-4. Epub 2019 Feb 1. PMID 30707299
- [Background] Finotto S, Bertolini G, Camellini R, Fantelli R, Formisano D, Macchioni MG, Mecugni D. Linguistic-cultural validation of the oral health assessment tool (OHAT) for the Italian context. BMC Nurs. 2020 Jan 31;19:7. doi: 10.1186/s12912-020-0399-y. eCollection 2020. PMID 32021562
- [Background] Ferrillo M, Migliario M, Roccuzzo A, Molinero-Mourelle P, Falcicchio G, Umano GR, Pezzotti F, Foglio Bonda PL, Calafiore D, de Sire A. Periodontal Disease and Vitamin D Deficiency in Pregnant Women: Which Correlation with Preterm and Low-Weight Birth? J Clin Med. 2021 Oct 2;10(19):4578. doi: 10.3390/jcm10194578. PMID 34640596
- [Background] Des Jarlais DC, Lyles C, Crepaz N; TREND Group. Improving the reporting quality of nonrandomized evaluations of behavioral and public health interventions: the TREND statement. Am J Public Health. 2004 Mar;94(3):361-6. doi: 10.2105/ajph.94.3.361. PMID 14998794
- [Background] Chalmers, J., Spencer, A., Carter, K., King, P., & Wright, C. (2009). Caring for oral health in Australian residential care. Dental Statistics and Research Series(48).
- [Background] Chalmers JM, King PL, Spencer AJ, Wright FA, Carter KD. The oral health assessment tool--validity and reliability. Aust Dent J. 2005 Sep;50(3):191-9. doi: 10.1111/j.1834-7819.2005.tb00360.x. PMID 16238218
- [Background] CDC. (2020, Aug. 28). CDC Oral Health. Retrieved Nov. 2020, from CDC Centers for Disease Control and Prevention: https://www.cdc.gov/
- [Background] Bhapkar, V. (1966, Mar.). A Note on the Equivalence of Two Test Criteria for Hypotheses in Categorical Data. Journal of the American Statistical Association, 61(313), 228-235. https://doi.org/10.2307/2283057.
- [Background] Ausserhofer D, Zander B, Busse R, Schubert M, De Geest S, Rafferty AM, Ball J, Scott A, Kinnunen J, Heinen M, Sjetne IS, Moreno-Casbas T, Kozka M, Lindqvist R, Diomidous M, Bruyneel L, Sermeus W, Aiken LH, Schwendimann R; RN4CAST consortium. Prevalence, patterns and predictors of nursing care left undone in European hospitals: results from the multicountry cross-sectional RN4CAST study. BMJ Qual Saf. 2014 Feb;23(2):126-35. doi: 10.1136/bmjqs-2013-002318. Epub 2013 Nov 10. PMID 24214796
- [Background] Arts DL, Voncken AG, Medlock S, Abu-Hanna A, van Weert HC. Reasons for intentional guideline non-adherence: A systematic review. Int J Med Inform. 2016 May;89:55-62. doi: 10.1016/j.ijmedinf.2016.02.009. Epub 2016 Feb 23. PMID 26980359
- [Background] Albrecht M, Kupfer R, Reissmann DR, Muhlhauser I, Kopke S. Oral health educational interventions for nursing home staff and residents. Cochrane Database Syst Rev. 2016 Sep 30;9(9):CD010535. doi: 10.1002/14651858.CD010535.pub2. PMID 27689868
- See also: CDC Oral Health. — https://www.cdc.gov/
- See also: Oral health for adults in care homes — https://www.nice.org.uk/guidance/ng48
- See also: Oral health: local authorities and partners — https://www.nice.org.uk/guidance/ph55
- See also: Oral health promotion in the community — https://www.nice.org.uk/guidance/qs139
- See also: RNAO. Best practice guidelines: oral health supporting adults — https://rnao.ca/bpg/guidelines/oral-health-supporting-adults-who-require-assistance-second-edition
- See also: World Health Organization. Health topics/Oral health — https://www.who.int/health-topics/oral-health/#tab=tab_1